CLINICAL TRIAL: NCT00675727
Title: Open Label, Single Arm, Phase I/II Study of CADI-05 in Patients With Advanced Stage III or Stage IV Melanoma
Brief Title: Safety Study of CADI-05 in Patients With Advanced Stage Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: DSMB reviewed data of 1st 10 subjects; determined no safety concerns. Efficacy as a single agent in this patient population was unlikely. Voluntary Termination
Sponsor: Cadila Pharnmaceuticals (Industry)
Responsible Party: Dr. Bakulesh M. Khamar, Director of Research, Cadila Pharmaceuticals Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-60/4051
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Stage III or Stage IV Melanoma
Keywords: Melanoma; Mycobacterium w
MeSH Terms: conditions — Melanoma | interventions — Immuvac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: CADI-05 — Two intradermal treatments each week for first 4 weeks followed by one intradermal treatment per week for second 4 weeks.

SUMMARY:
This study examines the safety of treating patients with advanced stage melanoma with the vaccine CADI-05. In addition, preliminary data regarding the clinical response and immune response will be collected.

DETAILED DESCRIPTION:
Because there are no highly effective treatment options for patients with advanced, unresectable melanoma, participation in clinical trials of novel therapies is frequently the best therapeutic alternative. CADI-05 is a promising agent for two reasons. First, patients with advanced melanoma frequently have disturbing symptoms such as anorexia with associated weight loss, fatigue, and chemotherapy-associated side effects such as nausea and vomiting. CADI-05 not only has a very low side effect profile, but it actually improves such symptoms. Second, melanomas are generally immunogenic, and sometimes patients mount significant of immune responses to cause spontaneous regression of tumors. High-dose interleukin-2, a relatively toxic therapy that stimulates the immune system, causes long-term regression in stage IV melanoma in a small percentage of patients. In addition, when combined with adoptive immunotherapy, response rates as high as 50% have been observed. Therefore, induction of potent antitumor immune responses in melanoma can be a highly effective therapeutic modality. Because CADI-05 has potent immunostimulatory effects and an excellent side effect profile, it is a very attractive option for treatment of stage IV melanoma patients. Preliminary data from ongoing preclinical studies in a murine melanoma model have shown that CADI-05 has significant biological activity in metastatic melanoma (G. Robertson, unpublished data).

Although it is possible that CADI-05 as a single agent will have activity in advanced melanoma, it may also be useful in conjunction with other systemic agents or as an adjuvant in conjunction with immunotherapy regimens. In addition, previous human trials suggest that CADI-05 may be helpful in symptom control and improvement of quality of life in patients with advanced melanoma. In spite of the promising data from a number of preclinical and clinical studies of this agent, no U.S. studies of the effects of CADI-05 in cancer patients have been performed. Therefore, the present research study proposes to evaluate the safety of CADI-05 treatment in advanced melanoma. In addition, preliminary data regarding the clinical response rate and immune response will be collected.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to understand and the willingness to sign a written informed consent document
* Subject must have a pathologic diagnosis malignant melanoma (stage III or IV).
* Subject must have at least one of the following:

  1. Melanoma that was previously treated with at least one complete or partial course of therapy for melanoma with either a poor to no response or evidence of disease progression;
  2. Melanoma that cannot be treated with first-line therapies because of medical comorbidities/risk of toxicity; or
  3. Melanoma that has not been treated with first-line therapies because of patient refusal.
* If melanoma is possibly resectable, the melanoma must have recurred despite at least two attempts at resection.
* The subject must have measurable disease, as defined by the presence of at least one measurable lesion, defined as having longest diameter greater than or equal to 20 mm by conventional measurement techniques (e.g., measurement of evaluable cutaneous metastases) or greater than or equal to 20 mm by imaging studies.
* Subject must have an ECOG performance status of 0, 1, or 2.
* Subject must have the ability to understand and provide informed consent that fulfills Institutional Review Board guidelines. Alternatively, if the subject is mentally incompetent for medical decision-making, a parent, legal guardian, or power of attorney has the ability to understand and provide informed consent that fulfills Institutional Review Board guidelines.
* Subject must be able to comply with office visits as required by the protocol.
* The effects of Investigational product on the developing human fetus is at the recommended therapeutic dose are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Subjects with medical co-morbidities, which in the judgment of the investigator, place them at an unacceptable level of risk for participation in this study.
* Pregnant women, since the prenatal effects of CADI-05 have not been characterized.
* Subjects with HIV, AIDS, or chronic immunosuppression for organ transplantation.
* Subjects who are unable to comply with office visits as required by this protocol or would suffer great hardship by participating in the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study.
* Clinically significant active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Recording of any clinical adverse reactions at anytime during the study for assessment of safety. | 6-24 months

SECONDARY OUTCOMES:
Both physical examinations and imaging studies will be used to evaluate clinical response to CADI-05 treatment. | 6-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Mosca, M.D., Ph.D., Principal Investigator — Lehigh Valley Hospital
Locations (1):
- Lehigh Valley Hospital, Allentown, Pennsylvania, United States